CLINICAL TRIAL: NCT01752842
Title: Lipid Biomarkers for Diabetic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Leducq Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201112122; P20HL113444-01 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Type II Diabetes Mellitus; Diabetes Complications
Keywords: Diabetes; Diabetic Cardiomyopathy; Triglycerides
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Diabetes Mellitus; Diabetic Cardiomyopathies | interventions — Fenofibrate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fenofibrate (Experimental): One fenofibrate 160 mg capsule per day for 12 weeks
  Interventions: Drug: Fenofibrate
- Placebo for fenofibrate (Placebo Comparator): One inert sugar pill per day for 12 weeks
  Interventions: Drug: Placebo for fenofibrate

INTERVENTIONS:
Drug: Fenofibrate
  Other Names: Tricor; Triglide; Antara; Lipofen
  Arms: Fenofibrate
Drug: Placebo for fenofibrate
  Other Names: Sugar pill manufactured to mimic Fenofibrate 160 mg capsule
  Arms: Placebo for fenofibrate

SUMMARY:
This study will test whether lowering the delivery of excess fats to the heart in persons with type-2 diabetes mellitus improves heart muscle function. The investigators will also test whether specific lipid molecular species in plasma can serve as biomarkers for diabetic heart disease.

DETAILED DESCRIPTION:
Screening procedures include 12-hour fasting blood draw, urine pregnancy testing for females, completion of medical history questionnaire, and stress echocardiography to rule out coronary artery disease or cardiomyopathy.

Subjects who meet screening criteria will return for visit 2, which consists of a urine collection, 12-hour fasting blood draw, dual-energy X-ray absorptiometry (DXA) for body composition, magnetic resonance spectroscopy analysis of the liver, and resting echocardiogram for analysis of heart structure and function. Subjects will then be randomized to treatment with fenofibrate (160 mg/d) or an identical-appearing placebo for 12 weeks. They will be asked to continue their usual medications, diet and physical activity. Subjects will receive a pedometer to wear daily to track their physical activity. Subjects will meet with dietitians from the Lifestyle Intervention Core to complete a 24-hour dietary recall. They will be instructed to record their daily blood glucose concentrations, distance walked and any side effects, illnesses or stresses in a study-supplied log. Subjects will be instructed to either email or fax the log to the study coordinator each week (or discuss by phone).

Subjects will return 6 weeks after starting intervention for visit 3 to ensure their medical safety. Procedures at this visit include an interim medical history, urine pregnancy test for females, blood draw to rule out untoward effects of the study drug on liver or kidney function, pill count to assess compliance, review of logs of blood glucose, distance walked, and side effects, illnesses or stresses, and meeting with a dietitian for a 24-hour dietary recall.

Subjects will continue to take their study medication/placebo and keep logs of blood glucose levels, distance walked, and side effects, illnesses and stresses for another 6 weeks. They will return for visit 4 after 12 total weeks of intervention. Visit 4 involves a urine collection, 12-hour fasting blood draw, review of subject logs, pill count, and 24-hour dietary recall. In addition, magnetic resonance spectroscopy analysis of the liver and resting echocardiogram analysis of the heart will be performed to determine if there have been any changes in liver fat or heart function during the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* body weight > 300 lb.
* HIV
* hypothyroid
* steroid medication, fenofibrate
* smoking
* BP > 140/90
* heart disease
* pregnant or lactating
* consumption of > 5 alcoholic drinks/wk
* creatinine > 1.5 mg/dL
* hematocrit < 28

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-03; Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean E Schaffer, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kannel WB, Hjortland M, Castelli WP. Role of diabetes in congestive heart failure: the Framingham study. Am J Cardiol. 1974 Jul;34(1):29-34. doi: 10.1016/0002-9149(74)90089-7. No abstract available. PMID 4835750
- [Background] Hamby RI, Zoneraich S, Sherman L. Diabetic cardiomyopathy. JAMA. 1974 Sep 23;229(13):1749-54. No abstract available. PMID 4278055
- [Background] Peterson LR, Herrero P, Schechtman KB, Racette SB, Waggoner AD, Kisrieva-Ware Z, Dence C, Klein S, Marsala J, Meyer T, Gropler RJ. Effect of obesity and insulin resistance on myocardial substrate metabolism and efficiency in young women. Circulation. 2004 May 11;109(18):2191-6. doi: 10.1161/01.CIR.0000127959.28627.F8. Epub 2004 May 3. PMID 15123530
- [Background] Herrero P, Peterson LR, McGill JB, Matthew S, Lesniak D, Dence C, Gropler RJ. Increased myocardial fatty acid metabolism in patients with type 1 diabetes mellitus. J Am Coll Cardiol. 2006 Feb 7;47(3):598-604. doi: 10.1016/j.jacc.2005.09.030. Epub 2006 Jan 18. PMID 16458143
- [Background] Szczepaniak LS, Dobbins RL, Metzger GJ, Sartoni-D'Ambrosia G, Arbique D, Vongpatanasin W, Unger R, Victor RG. Myocardial triglycerides and systolic function in humans: in vivo evaluation by localized proton spectroscopy and cardiac imaging. Magn Reson Med. 2003 Mar;49(3):417-23. doi: 10.1002/mrm.10372. PMID 12594743
- [Background] Sharma S, Adrogue JV, Golfman L, Uray I, Lemm J, Youker K, Noon GP, Frazier OH, Taegtmeyer H. Intramyocardial lipid accumulation in the failing human heart resembles the lipotoxic rat heart. FASEB J. 2004 Nov;18(14):1692-700. doi: 10.1096/fj.04-2263com. PMID 15522914
- [Background] Griffin JA, Osborn BW, Smithline HA. The impact of diabetes on hospital admissions, length of stay and mortality in emergency department patients with acute decompensated heart failure without ischemia. Acad Emerg Med. 2005;12:s97

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from clinics, practices and laboratories within the Barnes-Jewish Hospital consortium, Volunteer for Health and Diabetes Research Connections recruitment programs at Washington University School of Medicine, and through local advertisements, posters, emails and flyers. Dates of recruitment were from May 2013 to October 2017.
Pre-assignment Details: Potential subjects were given the approved consent form to consider. If interested, they were scheduled for a screening visit in the Center for Applied Research Sciences. The consent form was signed before any testing took place. Blood and urine were collected and a cardiac stress test was performed to evaluate the subject for eligibility.
Groups:
- Fenofibrate: Participants were instructed to take one fenofibrate 160 mg capsule every day for 12 weeks
  Fenofibrate
- Placebo for Fenofibrate: Participants were instructed to take one inert sugar pill every day for 12 weeks
  Placebo for fenofibrate
Period: Overall Study
Arm/Group | Fenofibrate | Placebo for Fenofibrate
Started | 34 | 36
Completed | 31 | 34
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Fenofibrate: One fenofibrate 160 mg capsule per day for 12 weeks
  Fenofibrate
- Placebo for Fenofibrate: One inert sugar pill per day for 12 weeks
  Placebo for fenofibrate
- Total: Total of all reporting groups
Arm/Group | Fenofibrate | Placebo for Fenofibrate | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (8.2) | 54.6 (8.3) | 54.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 27 | 26 | 53
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 36 | 70
Cardiac Diastolic Function (E') [Mean (Standard Deviation); unit: cm/s] — Population: Study-specific baseline characteristics were determined for subjects who completed the 12-week intervention only.
  cm/s
    number analyzed (Participants) | 31 | 34 | 65
    (all) | 8.30 (1.70) | 7.99 (1.78) | 8.1 (1.7)
Cardiac Systolic Function (Fractional Shortening) [Mean (Standard Deviation); unit: percent] — Population: Study-specific baseline characteristics were determined for subjects who completed the 12-week intervention only.
  percent
    number analyzed (Participants) | 31 | 34 | 65
    (all) | 39 (7) | 38 (6) | 38.2 (6.7)
C24:0/C16:0 ceramides [Mean (Standard Deviation); unit: ratio] — Population: Study-specific baseline characteristics were determined for subjects who completed the 12-week intervention only.
  ratio
    number analyzed (Participants) | 31 | 34 | 65
    (all) | 11.2 (2.4) | 12.4 (3) | 11.8 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Diastolic Function as Measured by E' (cm/s)
Description: Change was measured by echocardiography and was calculated as the value at 12 weeks minus the value at baseline.
Time Frame: Baseline and 12 weeks
Population: All participants for whom E' (diastolic function) was measured at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Fenofibrate | Placebo for Fenofibrate
Number analyzed (Participants) | 31 | 34
cm/s | -0.02 (1.35) | 0.55 (1.58)
Statistical Analysis 1: Comparison: Fenofibrate vs Placebo for Fenofibrate; Null hypothesis is no difference of mean change of cardiac diastolic function as measured by E' (cm/s) between placebo and Fenofibrate; Test type: Superiority — Power calculation is based on assumption that treatment with Fenofibrate will lead to 11% decrease in plasma TG and ceramide biomarkers. We also assume that there will be no significant change in ceramides without intervention. Based on these assumptions, 86 subjects are required to have 90% chance of detecting a decrease in the primary outcome measure from 1.29 in the placebo group to 1.15 in the Fenofibrate group; p = 0.07, ANCOVA — This P-value is based on ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.56 to 0.04] — ANCOVA was used to compare mean change of cardiac diastolic function adjusting for body fat percent, baseline values of BMI, diastolic/systolic blood pressure, HbA1c, fasting glucose, triglycerides, ethnicity, gender and race; Two-sample t-test was used to compare baseline mean values of biomarkers. All statistical tests are two-sided at significance level 0.05

2. Primary Outcome: Change in Cardiac Systolic Function as Measured by Fractional Shortening Percent
Description: Change was measured by echocardiography and was calculated as the value at 12 weeks minus the value at baseline.
Time Frame: Baseline and 12 weeks
Population: All participants for whom fractional shortening was measured at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Fenofibrate | Placebo for Fenofibrate
Number analyzed (Participants) | 31 | 34
percent | 0.025 (0.090) | 0.030 (0.083)
Statistical Analysis 1: Comparison: Fenofibrate vs Placebo for Fenofibrate; Null hypothesis is no difference of mean change of fractional shortening percent between placebo and Fenofibrate; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8128, ANCOVA — This P-value is based on ANCOVA; Mean Difference (Final Values) = 0.0058, 95% CI 2-sided [-0.0418 to 0.0543] — ANCOVA was used to compare mean change of outcome adjusting for body fat percent, demographic variables and baseline biomarkers; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Change in C24:0/C16:0 Ceramide Ratio
Description: Mass spectrometry-based quantification of the ratio of C24:0 ceramide to C16:0 ceramide in plasma.
Time Frame: Baseline and 12 weeks
Population: All participants for whom C24:0 and C16:0 ceramides were measured at baseline and 12 weeks.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fenofibrate | Placebo for Fenofibrate
Number analyzed (Participants) | 31 | 34
ratio | -1.6 (1.66) | -0.03 (2.44)
Statistical Analysis 1: Comparison: Fenofibrate vs Placebo for Fenofibrate; Null hypothesis is no difference of mean change of C24:0/C16:0 ceramide ratio between placebo and Fenofibrate; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0034, ANCOVA — This P-value is based on ANCOVA; ANCOVA was used to compare mean change of outcome adjusting for body fat percent, demographic variables and baseline biomarkers; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-2.93 to -0.65]; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 12 weeks of intervention.
Description: Participants self-reported side-effects weekly during intervention, and an interim study visit took place half-way through the 12 weeks so safety labs could be obtained.
Arm/Group | Fenofibrate | Placebo for Fenofibrate
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 2/34 | 0/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate (N=34) | Placebo for Fenofibrate (N=36)
rash/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Findings of this study cannot be extended to those who do not fit the entry criteria. Also, since this was a targeted lipidomics study, there may be changes in other lipid species after treatment with fenofibrate that were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT01752842/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT01752842/SAP_001.pdf